CLINICAL TRIAL: NCT02370706
Title: A Phase Ib, Multi-center, Open-label, Dose-escalation Study of PIM447 in Combination With Ruxolitinib (INC424) and LEE011 Administered Orally in Patients With Myelofibrosis
Brief Title: Study of the Safety of PIM447 in Combination With Ruxolitinib (INC424) and LEE011 in Patients With Myelofibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPIM447X2104C; 2014-003801-14 (EudraCT Number)
Record Dates: First submitted 2015-02-06; First posted 2015-02-25 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Myelofibrosis
Keywords: PIM447; LGH447; PIM inhibitor; LEE011; CDK 4/6 inhibitor; ruxolitinib; INC424; Jakavi®; Jakafi®; INCB18424; JAK inhibitor; myelofibrosis; PMF; PPV-MF; PET-MF
MeSH Terms: conditions — Primary Myelofibrosis | interventions — LGH-447; ruxolitinib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Arm 1 (Experimental)
  Interventions: Drug: PIM447; Drug: Ruxolitinib
- Dose Escalation Arm 2 (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: LEE011
- Dose Escalation Arm 3 (Experimental)
  Interventions: Drug: PIM447; Drug: Ruxolitinib; Drug: LEE011
- Dose Expansion Arm 1 (Experimental)
  Interventions: Drug: PIM447; Drug: Ruxolitinib
- Dose Expansion Arm 2 (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: LEE011
- Dose Expansion Arm 3 (Experimental)
  Interventions: Drug: PIM447; Drug: Ruxolitinib; Drug: LEE011

INTERVENTIONS:
Drug: PIM447 — pan-pim inhibitor
  Arms: Dose Escalation Arm 1; Dose Escalation Arm 3; Dose Expansion Arm 1; Dose Expansion Arm 3
Drug: Ruxolitinib — JAK1/JAK2 inhibitor
Drug: LEE011 — CDK4/6 inhibitor
  Arms: Dose Escalation Arm 2; Dose Escalation Arm 3; Dose Expansion Arm 2; Dose Expansion Arm 3

SUMMARY:
This is a phase Ib study with the primary purpose is to estimate the MTD and/or RDE for the triple combination of PIM447, formerly LGH447, plus ruxolitinib and LEE011 as well as for the doublets, PIM447 plus ruxolitinib, and LEE011 plus ruxolitinib, in patients with myelofibrosis (MF). Each regimen will be assessed for safety, tolerability, pharmacokinetics (PK) and pharmacodynamic effects, and preliminary anti-myelofibrosis activity, including changes in spleen volume, JAK2V617F allele burden, and hematologic response.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Patient must be diagnosed with JAK2V617F-positive primary or secondary MF.
* Dose-escalation and Expansion parts: Patients with a < 35% reduction in spleen volume by MRI/CT or < 50% reduction in spleen size by physical exam, with or without corresponding symptomatic improvement, after at least 6 months of treatment with single agent ruxolitinib at an optimal dose level in line with the label recommendations. Expansion parts only: Ruxolitinib-naive patients and patients who have been previously treated with single agent ruxolitinib and are relapsed and/or refractory.
* Patients must have splenomegaly measuring at least 5 cm by MRI at baseline.
* Have adequate bone marrow function:

  * Platelets ≥ 100,000 mm3 without the assistance of growth factors or platelet transfusions
  * Absolute Neutrophil Count (ANC) ≥ 1500/mm3 without growth factor support within 7 days prior to testing
  * Hemoglobin ≥ 9 g/dL.

Exclusion Criteria:

* Systemic antineoplastic therapy (including unconjugated therapeutic antibodies, toxin immunoconjugates, and alpha-interferon) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of study treatment
* Major surgery within 2 weeks before the first dose of either study drug.
* Patients who have had splenic irradiation within 2 weeks prior to Screening or prior splenectomy.
* Patients with AML, MDS, or peripheral blasts ≥ 10 %
* Prior autologous or allogeneic stem cell transplant at any time.
* Patients who are currently receiving treatment with a prohibited medication that cannot be discontinued at least one week prior to the start of treatment:

  * substrates of CYP3A4/5, CYP2B6 or CYP2D6 that have a narrow therapeutic window
  * strong inhibitors of CYP3A4/5 or CYP2D6
  * potent inducers of CYP3A4/5 or CYP2D6
* Serum total bilirubin > 1.5 x upper limit of normal (ULN) except in patients with Gilbert's syndrome who are excluded if the total bilirubin is > 3.0 x ULN or direct bilirubin > 1.5 x ULN, or aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or ALT (SGPT) > 3 x ULN, except in patients with MF involvement of the liver who are excluded if AST or ALT > 5 x ULN.
* Serum creatinine > 1.5 x ULN or calculated creatinine clearance < 60 ml/min according to Cockcroft-Gault equation
* Electrolyte abnormalities CTCAE grade ≥ 2 (e.g. serum potassium, magnesium and calcium) unless they can be repleted during screening and are deemed not clinically significant by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities during the first cycle of study treatment | Cycle 1 (28 days)
  To estimate the maximum tolerated dose and/or recommended dose for expansion for each of the following three treatment arms in patients with myelofibrosis (MF): PIM447 plus ruxolitinib (doublet), LEE011 plus ruxolitinib (doublet), PIM447 plus ruxolitinib and LEE 011 (triple combination).

SECONDARY OUTCOMES:
Number of participants with adverse events/serious adverse events | Approximately 27 months (end of study)
  Frequency and severity of adverse events (AEs), serious AEs (SAEs), changes in laboratory values, and electrocardiograms (ECGs), as a measure of safety and tolerability. Assessments consisted of recording all adverse events (AEs) and serious adverse events (SAEs), the regular monitoring of hematology, blood chemistry, urinalysis, and coagulation parameters, as well as electrocardiograms.
Proportion of patients achieving ≥ 35% reduction in spleen volume by magnetic resonance imaging (MRI) at Week 24 | 24 weeks
  To assess preliminary anti-myelofibrosis activity of PIM447 plus ruxolitinib, LEE011 plus ruxolitinib, and the triple combination PIM447 plus ruxolitinib and LEE011.
Changes in ratio of mutant to wild type JAK2 alleles (i.e. allele burden) | Approximately 27 months (end of study)
  To assess preliminary anti-myelofibrosis activity of PIM447 plus ruxolitinib, LEE011 plus ruxolitinib, and the triple combination PIM447 plus ruxolitinib and LEE011.
Change in platelets, neutrophils, and hemoglobin | Approximately 27 months (end of study)
  To assess preliminary anti-myelofibrosis activity of PIM447 plus ruxolitinib, LEE011 plus ruxolitinib, and the triple combination PIM447 plus ruxolitinib and LEE011.
Change in bone marrow fibrosis and histomorphology | Approximately 27 months (end of study)
  To assess preliminary anti-myelofibrosis activity of PIM447 plus ruxolitinib, LEE011 plus ruxolitinib, and the triple combination PIM447 plus ruxolitinib and LEE011.
Determine single and multiple dose pharmacokinetics (PK) profiles | Approximately 12 months
  Plasma concentration-time profiles of PIM447, ruxolitinib, and LEE011. PK parameters, including but not limited to Cmax, AUCinf, AUClast, AUCtau, T½, Tmax, accumulation ratio (Racc), CL/F, and Vz/F
Change in spleen volume as measured by MRI from baseline | Approximately 27 months (end of study)
  To assess preliminary anti-myelofibrosis activity of PIM447 plus ruxolitinib, LEE011 plus ruxolitinib, and the triple combination PIM447 plus ruxolitinib and LEE011.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, VIC, Melbourne, Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Villejuif, France
- Germany (2):
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Florence, FI, Italy
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CPIM447X2104C can be found on the Novartis Clinical Trial Results Website. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17874